CLINICAL TRIAL: NCT02210039
Title: Pilot Study to Image the Esophagus Using a SECM Probe
Brief Title: Using Spectrally Encoded Confocal Microscopy (SECM) to Visualise the Esophagus Using an SECM Probe
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Guillermo Tearney, Professor of Pathology, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 2013-P-001213
Record Dates: First submitted 2014-08-04; First posted 2014-08-06 (Estimated); Results first posted 2018-10-23 (Actual); Last update posted 2019-04-03 (Actual); Status verified 2019-04

CONDITIONS: Barrett's Esophagus
Keywords: SECM; Esophagus; Imaging
MeSH Terms: conditions — Barrett Esophagus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- SECM Probe Imaging (Experimental): SECM probe will be guided to a pre-determined length in the esophagus and spiral imaging will be performed using the SECM Imaging System.
  Interventions: Device: SECM Probe

INTERVENTIONS:
Device: SECM Probe — Imaging of the esophagus using SECM probe and system.

SUMMARY:
The study is being done to test the feasibility and tolerability of a SECM imaging probe in patients with Barrett's Esophagus (BE).

Subjects will undergo SECM probe imaging while they are under conscious sedation. Spiral SECM imaging will be performed continuously over a pre-determined length. Patients will later be asked for their feedback.

DETAILED DESCRIPTION:
Subjects with a previous diagnosis of Barrett's Esophagus will be recruited in the study and undergo SECM probe imaging while using conscious sedation, pulse oximetry and blood pressure monitoring. The probe will be inserted the predetermined required distance in the esophagus using a guide wire.

Once the SECM imaging probe is in place, spiral SECM image data will be continuously collected over a pre-determined length (approximately 5cm).

ELIGIBILITY:
Inclusion Criteria:

* A previous diagnosis of Barrett's Esophagus
* Patients must be over the age of 18
* Patient must be able to give informed consent

Exclusion Criteria:

* Subjects with any history of intestinal strictures
* OR subjects with a history of prior GI surgery
* OR subjects with a history of intestinal Crohn's disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2014-06; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Guillermo Tearney, MD, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | SECM Probe Imaging
Started | 6
Completed | 6
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | SECM Probe Imaging
Number analyzed (Participants) | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 4
  >=65 years | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.16 (12.20)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 6
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 6

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Tolerability of the Procedure
Description: We were monitoring the number of participants able to tolerate the procedure. All six participating subjects have been asked for a feedback about tolerability of the procedure using a specific tolerability questionnaire.
Time Frame: During the procedure
Population: All six study participants completed the study and the obtained data has been analyzed
Measure: Count of Participants; unit: Participants
Arm/Group | SECM Probe Imaging
Number analyzed (Participants) | 6
Participants | 6

ADVERSE EVENTS:
Time Frame: During the procedure
Description: The adverse events were collected systematically for this study. The definition of adverse events is the same as clinicaltrials.gov definition.
Groups:
- SECM Probe Imaging: SECM probe will be guided to a pre-determined length in the esophagus and spiral imaging will be performed using the SECM Imaging System.
  SECM Probe: Imaging of the esophagus using SECM probe and system.
  No adverse events has been reported.
Arm/Group | SECM Probe Imaging
All-Cause Mortality (participants affected / at risk) | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6
Other Adverse Events (participants affected / at risk) | 0/6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No